CLINICAL TRIAL: NCT01555723
Title: HIV (Human Immunodeficiency Virus) Subtype and ARV Response in African Children
Brief Title: Observational Study of Antiretroviral (ARV) Response in a Cohort of African Children Using Viral Load Monitoring
Acronym: RELATES
Status: Withdrawn | Type: Observational
Why Stopped: New study created.
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: RELATES
Record Dates: First submitted 2008-06-02; First posted 2012-03-15 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma obtained fron participants
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Treatment of HIV-1 infected Ugandan children with antiretroviral therapy (ART) is increasing but few prospective long-term studies evaluating the treatment process have been reported. In this study we sought to determine prospectively how consistent monitoring of HIV-1 RNA levels impacts the ART treatment process.

Methods: One hundred and eight children initiating ART were enrolled into this study. These children had comprehensive laboratory monitoring including HIV-1 RNA level determination and genotype analysis (where appropriate), CD4 % plus absolute counts, and safety laboratory measurements performed prior to starting therapy and at regular intervals after receiving ART. Kaplan-Meier statistics were used to examine predictors of survival and virologic failure. Viral genotype analysis was performed on samples obtained from children having virologic failure to determent the emergence of mutations.

DETAILED DESCRIPTION:
Study Setting The study was carried out at the Paediatric Infectious Disease Clinic (PIDC) now Baylor College of Medicine Bristol Myers Squibb Children's Clinical Centre of Excellence at Mulago Hospital. The PIDC is an HIV outpatient clinic operating 5 days a week with three paediatric clinics, one adolescent and one family-based clinic. The clinic provides care to one hundred and eighty children with HIV/AIDS daily. Approximately 50 children per month qualify for antiretroviral therapy based upon clinical and laboratory parameters.

The Makerere University Faculty of Medicine, Research Committee and Ethics Committee, the Uganda National Council of Science and Technology and IRB boards of Baylor College of Medicine and the University of Wisconsin Hospital and Clinics approved this study. Informed consent and assent (when applicable) was obtained from the primary caregiver and/or child before enrollment.

Study Participants and Enrollment Starting in 2007 children between the ages of 6 weeks and 18 years having confirmed HIV infection and receiving no ART were consecutively enrolled into this observational cohort study following consent and/or assent (where applicable). Children were excluded from participation if they were enrolled in another cohort study, or had psychosocial issues precluding participation (no parent or guardian willing to promote ART adherence or clinic HIV counselor evaluation of non adherence). The enrollment goal for this study was approximately100 children recruited over a period of 8 months.

Initiation of ART and Study Design Children confirmed to be HIV infected were screened with clinical history and examination by the study physician to determine eligibility. One hundred and twenty two children were recruited and 111 were enrolled into this prospective cohort study. Once enrolled a decision to start ART was based upon guidelines set forth by WHO (2006 guidelines with addendum in 2008)/UNAIDS recommendations, the Ugandan National Policy on ART and laboratory parameters (described below). ART treatment decisions were made at the discretion of the treating physician. Adherence monitoring was done by means of self-reporting and pill counts during patient visits to the clinic. Antiretroviral (ARV) medications used in the study included: zidovudine (AZT), lamivudine (3TC), abacavir (ABC), stavudine (d4T), nevirapine (NVP), efavirenz (EFV), didanosine (ddI), tenofovir/emtricitabine (Truvada), lopinavir/ritonavir (Aluvia/Kaletra). History of peripartum NVP use by the child and/or mother was obtained through interview.

Clinical assessment with disease staging (both WHO and CDC) and baseline laboratory investigations which included complete blood count (CBC), renal and liver function tests (RFT and LFT, respectively), CD4%/absolute count, HIV-1 RNA level and genotype were done prior to the patient starting ART. All blood samples were labeled with a study number that was used for participant identification. Clinical assessment was done at every patient visit. VL monitoring was done every three months during the first year of ART follow up and every 6 months thereafter to the end of the study period. CD4%/absolute count and safety laboratory evaluations were done every 6 months. Genotype evaluation was done prior to starting therapy and when virological failure was documented. Virologic failure was defined as two consecutive (for our clinic one month apart) HIV-1 RNA levels >400 copies/ml occurring at any time during the study period in a child who previously was suppressed or had a 1-2 log10 response to ART; a persistent viral load elevation (>400 copies/ml) during the first 3 months of ART; or a viral load >1000 copies/ml on the last blood drawn from a child at the end of the study period, before death, or at withdrawal or lost to follow-up. Initial virologic response was defined as a decrease in the HIV-1 RNA level (viral load) of at least 1 log from baseline after 4-8 weeks of ART. A full virologic response was defined as an HIV-1 RNA level <400 copies/ml (undetectable) by week 24 and/or 48 after starting ART.

Successful immunologic reconstitution was defined as an increase of at least 10 percentage points over the baseline CD4 percent level occurring within the first year of therapy. An absolute CD4 cell count response to ART was defined as an increase of 50-150 cells/mm3 over baseline levels occurring within the first year of therapy. A sustained decline of 5% in the CD4%, a decline below the pre-therapy CD4% or absolute count or no change in the baseline CD%/absolute count was used to define immunologic failure.

Laboratory Measurements Complete blood count (CBC), liver function (ALT), renal function (creatinine), CD4 percent/absolute count and plasma HIV-1 RNA were performed at the Makerere University-Johns Hopkins University (MU-JHU) core laboratory, Kampala, Uganda (certified by the College of American Pathologists). CD4%/ absolute counts were assessed using a BD FACS Calibur instrument (Becton, Dickinson and Company). The plasma HIV-1 RNA level was measured using the Amplicor HIV-1 Monitor Test Standard assay (version 1.5, Roche Company, Branchburg, NJ/USA). We report plasma HIV-1 RNA levels as log10 in this study.

HIV-1 subtyping and genotyping was assessed using the GeneSeq technique at Monogram Bioscience, South San Francisco CA/USA. In this assay, amplifying the pool of virus variants in the plasma sample using the polymerase chain reaction (adapted for use with non-subtype B virus) product enabled construct of resistance vector DNA pools. Deduced amino acid sequences and drug susceptibility of sample virus were compared with a reference virus strain to identify mutations. Genotype analysis was conducted only on blood samples having >1000 copies of virus particles per ml. The GeneSeq HIV assay detects minor virus populations at concentrations above 10-20%.

Statistical Analysis Survival and virologic treatment failure analyses were evaluated with Kaplan-Meier statistics. Cox Regression multivariate analysis and Kaplan-Meier statistics were used to examine the relationship of clinical and laboratory parameters to virologic failure and a t-test of significance was used to evaluate the immunologic (mean CD4 %/absolute count at different time points) response to ART.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 6 weeks and 18 years having confirmed HIV infection
* Receiving no ART were consecutively enrolled into this observational study
* Consent and/or assent (where applicable) had to be obtained.

Exclusion Criteria:

* Children were enrolled in another cohort study
* Had psychosocial issues precluding participation (no parent or guardian willing to promote ART adherence or clinic HIV counselor evaluation of non adherence).

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Inclusion Criteria: Starting in 2008 children between the ages of 6 weeks and 18 years having confirmed HIV infection and receiving no ART were consecutively enrolled into this observational cohort study following consent and/or assent (where applicable).
  Exclusion Criteria: Children were excluded from participation if they were enrolled in another cohort study, or had psychosocial issues precluding participation (no parent or guardian willing to promote ART adherence or clinic HIV counselor evaluation of non adherence). The enrollment goal for this study was approximately100 children recruited over a period of 8 months.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank M Graziano, MD PhD, Principal Investigator — U Wisconsin